CLINICAL TRIAL: NCT06446557
Title: De-scalation or swItch of Treatment According to Circulating tuMOr DNA Variation After 2 Cycles of Doublet Chemotherapy Plus Targeted Agent in Metastatic Unresectable Colorectal Cancer (DIAMOND Study): A Randomized Phase III of PRODIGE Intergroup
Brief Title: De-scalation or swItch of Treatment According to Circulating tuMOr DNA Variation After 2 Cycles of Doublet Chemotherapy Plus Targeted Agent in Metastatic Unresectable Colorectal Cancer
Acronym: DIAMOND
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/0343/HP
Record Dates: First submitted 2024-02-26; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): After 4 cycles of doublet + TA, non-progressive patients will be allocated to a strategy according to ctDNA value and variation from C1-C3
  Interventions: Drug: treatment adaptation guided by ctDNA variation
- Arm B (Active Comparator): At least 8 cycles of doublet CT + TA before adaptation of sequence at physician choice.
  Interventions: Drug: standard management

INTERVENTIONS:
Drug: treatment adaptation guided by ctDNA variation — after 4 cycles of doublet + TA, non-progressive patients will be allocated to a strategy according to ctDNA value and variation from C1-C3: Arm A1: CT discontinuation (ctDNA normalization < 0.1 ng/ml or ctDNA not detectable) Arm A2 : maintenance with fluoropyrimidine + TA (ctDNA ≥ 0.1 ng/ml and ∆ctDNA≥ 80%).
  Arm A3 : ctDNA non-responders (∆ctDNA < 80% or increase) : switch of CT +/- TA.
  Arms: Arm A
Drug: standard management — At least 8 cycles of doublet CT + TA before adaptation of sequence at physician choice.
  Arms: Arm B

SUMMARY:
Background : In unresectable mCRC, a de-escalation strategy using maintenance or chemotherapy (CT) discontinuation in selected cases is considered as a valid option in non-progressive patients after a first-line induction of doublet CT + targeted agent (TA) (1-7).

In this context, circulating tumor DNA (ctDNA) is considered very promising to optimize decision making. Indeed, ctDNA harbour the same main alterations of the tumor and has been recognized as biologically relevant to reflect tumor dynamics and therapeutic efficacy (8).

As we and other groups reported in mCRC, that early variation of ctDNA during CT may be relevant to predict outcome (9-11). Indeed, patients with a ctDNA decrease from the first (C1) to the third (C3) cycles of CT (∆≥80% or ctDNA<0.1 ng/ml at C3) or without ctDNA detectable at C1 and C3 have significant better survival as compared to patients with less decrease or with ctDNA increase (10). ctDNA monitoring had never been prospectively evaluated to guide early adaptation in the treatment strategy in mCRC.

Aim: A randomized phase III, open label, strategy trial of the superiority in overall survival (OS) adjusted on quality of life of an early treatment adaptation guided by ctDNA variation versus a standard management in unresectable left-side, MSS-BRAFV600E non-mutated mCRC treated by first-line doublet CT + TA.

Patients and methods :

-Main inclusion criteria will be (i) unresectable left-side and non-pre-treated mCRC (ii) MSS and non-mutated BRAFV600E tumor (iii) at least one measurable lesion (iv) ECOG 0-1 and adequate biological functions for first-line doublet CT + TA (antiEGFR if RAS WT, bevacizumab (BV) if RAS MUT).

Randomization (1:1) between an experimental strategy guided by ctDNA variation with de-escalation (Arm A1 or A2) or switch of treatment (Arm A3) versus standard strategy (Arm B). The analysis of variation of ctDNA from C1-C3 will be centralized and detected using Digital PCR targeting hypermethylation of WIF1/NPY genes (10) in real-time in arm A and in second step in arm B.

Randomization in Arm A: after 4 cycles of doublet + TA, non-progressive patients will be allocated to a strategy according to ctDNA value and variation from C1-C3:

Arm A1: CT discontinuation (ctDNA normalization < 0.1 ng/ml or ctDNA not detectable) Arm A2 : maintenance with fluoropyrimidine + TA (ctDNA ≥ 0.1 ng/ml and ∆ctDNA≥ 80%).

Arm A3 : ctDNA non-responders (∆ctDNA < 80% or increase) : switch of CT +/- TA.

Randomisation in Arm B: at least 8 cycles of doublet CT + TA before adaptation of sequence at physician choice.

Statistical considerations : with an expected median OS at 32 months (mean 37.6 months), a mean QoL at 70.0% in first-line mCRC, corresponding to 0.700 x 37.6 = 26.3 QALM or 2.19 QALY (SD 1.18 QALY), 408 patients are required (randomization 1:1) to show a gain of 4 months of quality-adjusted OS (4 QALM or 0.33 QALY) in experimental ctDNA strategy versus standard strategy (5% two-sided type I error rate, 81% power and 1.18 QALY SD).

The secondary objectives will be:

* To compare strategies (standard vs ctDNA guided) overall and in the subgroups of ctDNA response on 18, 24 and 36-months restricted mean of QoL-adjusted OS, OS, PFS, response rate, toxicity, Quality of Life and cost utility.
* Bio-collection for further ctDNA analysis. Only cost of samples collection and their transportation to the resource center is requested. Further ancillary analysis will be subject to independent funding requests to evaluate :
* ctDNA kinetics during the induction and its impact on outcome in overall population and in each arm
* ctDNA changes between time points during de-escalation arms to determine thresholds of variations predictive of clinical and/or radiological progression.

Conclusion: DIAMOND is a randomized phase III strategy trial to show the superiority in OS adjusted on quality of life of an early treatment adaptation guided by ctDNA versus a standard management in unresectable left-side, MSS-BRAFV600E non-mutated mCRC treated by first-line doublet CT + TA.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of RAS WT or mutant, MSS, BRAFV600E non-mutated colorectal cancer.
* Left side or rectal cancer
* An unresectable metastatic colorectal cancer not previously treated with chemotherapy for metastatic disease.
* At least one measurable lesion according to RECIST criteria version 1.1.
* Age ≥ 18 years.
* ECOG PS ≤ 1
* Neutrophils ≥ 1.5 x 10^9/L, Platelets ≥ 100 x 10^9/L, Hb > 9 g/dl.
* Total bilirubin ≤ 1.5 time the upper-normal limits (UNL) and ASAT (SGOT) and/or ALAT (SGPT) ≤ 2.5 x UNL, or 5 x UNL in case of liver metastases, alkaline phosphatase ≤ 2.5 x UNL, or 5 x UNL in case of liver metastases.
* Creatinine clearance > 50 mL/min or serum creatinine ≤ 1.5 x UNL.
* The patient's urinary protein is ≤ 1+ on dipstick or routine urinalysis.
* Adequate coagulation function [International Normalized Ratio (INR) ≤1.5 and Partial. Thromboplastin Time (PTT) or activated PTT (aPTT) ≤1.5 x ULN.
* Written informed consent.

Exclusion Criteria:

* Right side colon cancer
* First-line chemotherapy +/- biologic agents for mCRC before C1
* Radiotherapy to any site within 4 weeks before C1
* Adjuvant oxaliplatin-based treatment completed less than 6 months before relapse.
* Treatment with any investigational drug within 30 days prior to C1
* Known allergy to any of the study treatment components.
* Dihydropyrimidine dehydrogenase (DPD) deficiency.
* Documented and/or symptomatic brain or leptomeningeal metastases.
* Patient with active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia, uncontrolled thrombotic or hemorrhagic disorder, or any other serious uncontrolled medical disorders in the opinion of the investigator.
* Uncontrolled or poorly controlled hypertension despite standard medical management.
* Severe renal or hepatic failure
* Serious or non-healing wound, ulcer, or bone fracture within 28 days prior to C1
* Other co-existing malignancies or malignancies diagnosed within the last 3 years with the exception of basal and squamous cell carcinoma or cervical cancer in situ.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start.
* Infection with the human immunodeficiency virus.
* Symptomatic peripheral neuropathy grade 1 according the NCI CTC.
* Acute or subacute bowel obstruction or history of chronic diarrhea, which is considered clinically significant in the opinion of the investigator.
* Chronic antiplatelet therapy, including aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted.
* Pregnant or lactating women.
* Patient with active psychiatric illness or social situation that would severely limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the superiority in quality-adjusted OS of an early treatment adaptation guided by ctDNA variation | through study completion, an average of 7 years
  The primary endpoint is the superiority in overall survival (OS) adjusted on quality-adjusted life years (QALYs) for the experimental arm guided by ctDNA (Arm A1 + A2 + A3) as compared to the standard management (Arm B).
  The follow-up will start from the date of randomization. Patients alive at last follow-up will have an extrapolation of their QALY, based on the OS curve and the patient QoL at last follow-up.

IPD SHARING:
Plan to Share IPD: No